CLINICAL TRIAL: NCT01483469
Title: Human Proof of Concept Positron Emission Tomography Study to Investigate [11C]-RO5011232 as a Radiotracer for Brain mGlu5 Receptor Occupancy and to Investigate the Binding of RO4917523 to Human mGlu5 Brain Receptor at Steady-state.
Brief Title: A Human Proof of Concept Study for [11C]-RO5011232 as Radiotracer and Study of the Binding of RO4917523 to Human mGlu5 Brain Receptor at Steady-State in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: BP27890
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 2-chloro-4-(1-(4-fluorophenyl)-2,5-dimethyl-1H-imidazol-4-ylethynyl)pyridine

ARMS (2):
- Concept Proof (Active Comparator)
  Interventions: Drug: RO5011232
- Receptor Occupancy (Experimental)
  Interventions: Drug: RO4917523; Drug: RO5011232

INTERVENTIONS:
Drug: RO4917523 — orally daily, 14 days
  Arms: Receptor Occupancy
Drug: RO5011232 — [11C]-RO5011232 intravenously

SUMMARY:
This open label, non-randomized, parallel group study will evaluate [11C]-RO5011232 as radiotracer for brain mGlu5 receptor occupancy and investigate the binding of RO49917523 to human mGlu5 brain receptor at steady-state in healthy volunteers. In Parts I, II and III, positron emission tomography (PET) assessments of specific uptake of the radiotracer and whole body dosimetry will be made after intravenous injection of [11C]-RO5011232. In Part IV, subjects will receive RO4917523 orally daily for 14 days while receiving three single intravenous bolus injections of [11C]-RO5011232. The anticipated time on study treatment is up to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers as determined by medical history, physical examination, 12-lead ECG, and routine clinical laboratory measurements
* Age 18 to 65 years inclusive
* Body mass index (BMI) between 18 to30 kg/m2 inclusive and body weight at least 50 kg
* Appropriate body size (less than 195 cm [6 feet and 5 inches]) in order to accommodate the whole body scanning

Exclusion Criteria:

* History of or presence of clinically significant psychiatric condition, as evaluated by a psychiatrist before enrolment
* History of head trauma with prolonged loss of consciousness (>10 minutes) or any neurological condition or a history of migraine headaches
* Contraindications to MRI procedures (Part I, III and IV)
* Subjects suffering from claustrophobia or who would be unable to undergo magnetic resonance imaging (MRI) or PET scanning
* Positive pregnancy test at screening or on any day preceding a PET scan
* Lactating women
* Positive for hepatitis B, hepatitis C or HIV infection
* Any history of alcohol or drug abuse within the last 6 months
* Regular smoker or nicotine user (>10 cigarettes per day)
* Participation in an investigational drug or device study within three months prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Part I: mGlu5 receptor binding of [11C]-RO5011232 radiotracer in human brain, assessed by positron emission tomography (PET) | approximately 6 months
Part II: Dosimetry/radiation safety of [11C]-RO5011232 assessments by whole body PET scan | approximately 6 months
Part III: Measurement of test-retest precision of PET images of regions of interest in the human brain | approximately 6 months
Part IV: Correlation between RO4917523 plasma concentration and R04917523 binding to mGlu5 receptor in brain | approximately 6 months

SECONDARY OUTCOMES:
Safety of [11C]-RO5011232 administered intravenously at microdose level: Incidence of adverse events | approximately 6 months
Part IV: In vitro binding potential (reference region with no specific binding of radiotracer) assessed by PET | approximately 6 months
Part IV: Safety of 14-day treatment with RO4917523: Incidence of adverse events | approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Baltimore, Maryland, United States